CLINICAL TRIAL: NCT01672840
Title: Effects of Cocoa on Ambulatory Blood Pressure and Vascular Function in Patients With Stage I Hypertension
Acronym: DARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-03
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Stage 1 Hypertension; cocoa consumption; Blood pressure; Endothelial function; arterial stiffness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5g Cocoa Consumption (Experimental): Daily consumption of 10g Extra Dark cholocate and a beverage containing 2.5g of cocoa powder for 8 weeks
  Interventions: Dietary Supplement: 5g Cocoa Consumption
- 10g Cocoa Consumption (Experimental): Daily consumption of 20g Extra Dark cholocate and two beverage containing 2.5g of cocoa powder each for 8 weeks
  Interventions: Dietary Supplement: 10g Cocoa Consumption

INTERVENTIONS:
Dietary Supplement: 5g Cocoa Consumption — Daily consumption of 10g Extra Dark cholocate and a beverage containing 2.5g of cocoa powder for 8 weeks
  Arms: 5g Cocoa Consumption
Dietary Supplement: 10g Cocoa Consumption — Daily consumption of 20g Extra Dark cholocate and two beverage containing 2.5g of cocoa powder each for 8 weeks
  Arms: 10g Cocoa Consumption

SUMMARY:
The proposed study Dose And Response to Cocoa (DARC), will examine variation in dose of cocoa-containing product consumption over an 8-week period and assess effects on blood pressure, endothelial function and arterial stiffness. The randomized, controlled, modified Latin square parallel design will compare the effects of two doses of cocoa consumption on blood pressure, endothelial function and arterial stiffness in 120 adults with stage 1 hypertension.

DETAILED DESCRIPTION:
Hypothesis #1 To verify the efficacy of an 8-week course of cocoa-containing product consumption on blood pressure in adults with stage 1 hypertension. Specifically, to demonstrate at least 3.5 mmHg improvement in 24-hour mean systolic blood pressure following 8 weeks of treatment with cocoa- containing products when compared to placebo. Our hypothesis is that cocoa-containing product consumption will result in clinically significant improvement of systolic blood pressure at the conclusion of an 8-week course of treatment.

Hypothesis #2 To identify a dose-response relationship in which increasingly higher doses of cocoa powder in cocoa-containing products will demonstrate correspondingly greater beneficial effects on blood pressure over an 8-week period in individuals with stage 1 hypertension. Specifically, to investigate the effects of the variation of dose of cocoa powder in cocoa-containing products (i.e. 5 grams or 10 grams of cocoa powder) for 8 weeks on blood pressure. We hypothesize that increasingly higher doses of cocoa powder in cocoa-containing products will demonstrate correspondingly greater beneficial effects on blood pressure.

Hypothesis #3 To assess the effects of different doses of cocoa-containing product consumption over an 8-week period on 24-hour diastolic blood pressure, endothelial function, arterial stiffness, serum lipids, theobromine, CRP, glucose, insulin, body weight, and waist circumference in adults with stage 1 hypertension. We hypothesize that consumption of cocoa-containing products will lower diastolic blood pressure; improve endothelial function of our participants; reduce arterial stiffness; improve serum lipids; theobromine; and will have no clinically meaningful effects on body weight and waist circumference, CRP, glucose, or insulin.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 18-75 years
* stage 1 hypertension (i.e. 140-159/90-99 mmHg) without anti-hypertensive medication or with only one anti-hypertensive medicaion
* body mass index < 35 kg/m²
* willing to discontinue the use of chocolate/cocoa products at least 4 weeks prior to intervention.

Exclusion Criteria:

* anticipated inability to complete or comply with study protocol
* use of lipid-lowering or aspirin unless stable on medication for at least 1 month and willing to refrain from taking medication for 12 hours prior to endothelial function scanning
* severe hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100 mmHg), or use more than one anti-hypertensive medications
* allergic to cocoa products (chocolate or cocoa powder)
* regular use of vitamin C, vitamin E, fish oil, flax seed oil, omega-3 fatty acids, Coenzyme Q10, fiber supplements, garlic pills, arginine, red yeast rice, and/or any kind of antioxidant and unwilling to discontinue supplementation for at least 4 weeks prior to study initiation and for the study duration. Use of a multi-vitamin containing no more than two times the recommended daily allowance for vitamins C and E is permissible
* diagnosed eating disorder
* on any specific diet, weight control diet, and/or vegan diet
* substance abuse (chronic alcoholism and/or other chemical dependency)
* any unstable medical condition that would limit the ability of a subject to participate fully in the trial (e.g., cancer, AIDS, tuberculosis, psychotic disorder)
* current or impending pregnancy. In premenopausal women, pregnancy will be excluded by pregnancy test at the time of each study visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring (ABPM) | 8 weeks
  Subjects will undergo 24-hour ambulatory blood pressure monitoring using a FDA approved device (Model 90207 with standard adult cuff or large cuff (depending on arm size), Spacelabs Medical, Inc.). BP will be measured every 30 minutes throughout the 24-hour monitoring period. Mean systolic, mean diastolic, and average mean blood pressure will be calculated from all valid BP measurements. Daytime and nighttime (11:00 PM till 6:30 AM) BP will also be assessed.
Office Blood Pressure | 8 Weeks
  Systolic and diastolic BP will be measured at each visit using an approved automated device. Blood pressure will be measured (average of three measurements with five minutes between measurements) with the participant sitting in a quiet room.

SECONDARY OUTCOMES:
Flow-mediated dilatation (FMD) | 8 Weeks
  FMD will be measured as the percent change in brachial artery diameter from pre-cuff inflation to 60-seconds post-cuff release (upper arm cuff position). In addition to brachial diameter at 60 seconds post-cuff release, flow after cuff deflation within the first 15 seconds will be used as an indicator of stimulus strength, hyperemic flow being the stimulus for endothelial reactivity.
Central Aortic Stiffness | 8 Weeks
  First, we will examine pulse pressure, which reflects central arterial stiffness and is an important predictor of cardiovascular disease mortality in hypertensive subjects. Then, we will use recently developed non-invasive methodology that examines carotid-femoral pulse wave velocity. Carotid femoral pulse wave velocity will be measured using the SphgymoCor (AtCor, Medical, Inc.). This measure will be assessed in a subgroup of the study population (n=50) at the University of Boston site.
Fasting Serum Lipids | 8 Weeks
  Total cholesterol (Tchol), triglycerides (TG), and high-density lipoprotein (HDL) will be obtained by direct measurements. Very-low-density lipoprotein (VLDL) and low-density-lipoprotein (LDL) will be obtained by calculation: VLDL = TG/5; and LDL = Tchol - (VLDL + HDL). HDL:Tchol ratio will be used to evaluate the impact of treatment assignments on lipid panel.
C-Reactive Protein (CRP) | 8 Weeks
  Serum CRP values will be determined using a high sensitivity CRP (hsCRP) ELISA method.
Fasting Glucose and Insulin | 8 Weeks
  Glucose and insulin will be measured at each time point. HOMA-IR will be calculated.
Body Weight | 8 Weeks
  Body weight will be measured for all study participants during each visit. Body weight will be measured to the nearest 0.5 pound using a balance-type medical scale. Subjects will be measured in the morning (fasting), unclothed with the exception of undergarments.
Waist Circumference | 8 Weeks
  Waist circumference will be measured using the U.S. government standard protocol. Waist circumference will be measured around the narrowest point between ribs and hips when viewed from the front after exhaling.
3- Day Food Diary | 8 Weeks
  Food diaries will be used to track any variation in the dietary pattern over the course of the study. The study coordinators will instruct participants on how to accurately complete a food diary, and will answer any questions posed by participants at the clinical screening. All participants will be asked to complete food diaries after clinical screening and at the end of each treatment assignment. Diet records will be analyzed by a registered dietitian using basic nutrition and diet analysis software (The Food Processor II, version 7.0; ESHA Research, Salem, OR).
Physical Activity | 8 Weeks
  Physical activity will be determined by the Seven-Day Physical Activity Recall [PAR]. The PAR provides detail regarding the duration, intensity, and volume (energy expenditure) of physical activity and can therefore be used for a variety of applications. Because it utilizes a one-week time frame, the data from the PAR is often considered representative of typical activity patterns. While it requires considerable cognitive effort by the participants, the interviewer administered version can be completed in a reasonable amount of time (~20 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Valentine Njike, MPH, MD, Principal Investigator — Yale-Griffin Prevention Research Center; Joseph A. Vita, MD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Griffin Hospital, Derby, Connecticut
  - Boston University School of Medicine, Boston, Massachusetts